CLINICAL TRIAL: NCT06054087
Title: Effectiveness of Electroacupuncture in the Treatment of Diabetic Peripheral Neuropathy: a MulticentreRandomised Controlled Trial
Brief Title: Effectiveness of Electroacupuncture in the Treatment of Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); The Second Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, professor, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GZY-ZJ-KJ-23021-01
Record Dates: First submitted 2023-09-05; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Diabetic Peripheral Neuropathy; Electroacupuncture; Multi-center RCT

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EA group (Experimental): Subjects in this group received electroacupuncture along with the basic treatment at a frequency of 2 treatments per week for 6 weeks for a total of 12 interventions. The follow-up period is one month.
  Interventions: Procedure: Basal therapy+EA
- Waiting list group (Other): The subjects in this group will receive only basal treatment with no additional therapies during the study period. After the end of the study period, patients were given 12 acupuncture treatments
  Interventions: Other: Basal therapy

INTERVENTIONS:
Procedure: Basal therapy+EA — 1. Participants are not set up with uniform medication. High blood sugar is controlled by hypoglycaemic drugs, patients with hypertension and hyperlipidaemia can take antihypertensive and lipid-lowering drugs, while other drugs are based on the patient's current medication.
  2. Main acupoints: Qihai (RN6), Guanyuan (RN4), Xuehai (SP10), Yanglingquan (GB34), Zusanli (T36), Yinlingquan (SP9), Sanyinjiao (SP6), Xuanzhong (GB39), Jiexi (ST41), Zulinqi (GB41), Taichong (SP41). Supporting acupoints: for pain in the upper limbs, add Baxie, Quchi (LI11), Shousanli (LI10), Hegu (LI4), and Ashixue; for pain in the lower limbs, add Bafeng, Neiting (ST44),Kunlun (BL60). Operation: Acupuncture needles of size 25*40mm will be used. The electrode will be connected Yanglingquan (GB34) and Sanyinjiao (SP6), electrode wire will be connected to the electro-acupuncture apparatus using continuous wave with a frequency of 2Hz at an intensity suitable for the comfort of the subject.
  Arms: EA group
Other: Basal therapy — Participants are not set up with uniform medication. High blood sugar is controlled by hypoglycaemic drugs, patients with hypertension and hyperlipidaemia can take antihypertensive and lipid-lowering drugs, while other drugs are based on the patient's current medication.
  Arms: Waiting list group

SUMMARY:
Diabetic Peripheral Neuropathy (DPN) is one of the most common chronic complications of diabetes mellitus, which mainly manifests symmetric pain, numbness, ankylosis, or with abdominal distension, abnormal sweating, and accompanied by glove-sock-like hyperalgesia or loss of sensation as the main symptom, which seriously affects the quality of life of patients. Although drug treatment has some effect, from the overall long-term perspective, long-term medication is easy to produce drug dependence, and often easy to cause ataxia, blurred vision, constipation, diplopia, nausea and other adverse drug reactions. Electroacupuncture treatment for DPN has certain advantages, with clear efficacy and no toxic side effects, and is being increasingly recognised by the public and professionals. The study is designed to observe the therapeutic effect and safety of electroacupuncture (EA) in the treatment of DPN.

DETAILED DESCRIPTION:
A total of 104 subjects with DPN who meet the inclusion criteria will be included in the study. Subjects will be classified as mild, moderate and severe in terms of severity by using the toronto clinical scoring system（TCSS）, and subsequently randomised into the EA group and the waiting list group by using a central randomisation system. The indexes of main outcome evaluation are: sensory nerve conduction velocity (SNCV) and motor nerve conduction velocity (MNCV) of the tibial and peroneal nerves of the lower extremities. The indexes of secondary outcome evaluation are: 1) Overall clinical effectiveness rate; 2) TCSS score; 3) Chinese medicine symptom score; 4) patient's global impression of change (PGIC); 5) regional temperature test; and 6) laboratory tests (glycosylated haemoglobin, fasting blood glucose, and postprandial 2h blood glucose). This study will evaluate the effectiveness of EA in treating DPN and assess the difference in the efficacy of EA in treating patients with DPN of different severity, as well as explore the feasibility of regional temperature as an indicator for assessing the efficacy of DPN. And based on the results, a standardised, effective and convenient EA treatment protocol will be established for promotion.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years ≤ age ≤ 85 years, disease duration is not limited, gender is not limited;
2. Lower limb neuromuscular electromyography showing reduced conduction velocity, and/or persistent pain and/or sensory abnormalities in the extremities (at least in both lower limbs), bilateral or unilateral weakened ankle reflexes, reduced vibration sensation, and a TCSS score ≥ 6;
3. Have normal communication skills;
4. No serious heart, brain, liver, kidney and other internal diseases, no serious mental illness and cognitive impairment;
5. those who voluntarily obeyed the study protocol and signed the informed consent form.

Exclusion Criteria:

1. Persons with peripheral neuropathy, ulcers and gangrene of the limbs caused by a variety of other reasons (e.g. hypothyroidism, alcohol, drugs, heredity, etc.), or persons with a history of skin ulcers or lesions that do not heal easily;
2. Presence of serious diseases, including renal disease, cardiovascular disease, pulmonary disease, liver disease or infectious disease, or malignant tumour and serious mental illness, etc;
3. Prior history of knee/hip replacement surgery or lower limb fracture within the past 3 months, and other conditions that may affect the assessment of neuropathy
4. Patients who have received acupuncture or moxibustion treatment for DPN within the past 3 months;
5. Volunteers who are participating in other interventional clinical trials;
6. Women who are preparing for pregnancy, pregnant or breastfeeding;
7. Those who have scars or hyperpigmentation of the skin at the testing site, which affects the accuracy of the test;
8. Unwilling to be randomly assigned to the waiting treatment group or electroacupuncture treatment group;
9. Chronic abuse of opioids, analgesics, illicit drugs or alcohol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensory conduction velocity of superficial peroneal nerve | Baseline, 6 weeks
Sensory conduction velocity of sural nerve | Baseline, 6 weeks
Motor conduction velocity of Peroneal nerve | Baseline, 6 weeks
Motor conduction velocity of tibial nerve | Baseline, 6 weeks

SECONDARY OUTCOMES:
Overall clinical effectiveness rate | 3 weeks, 6 weeks, 10 weeks
  Total effective rate = [(number of cured cases + number of effective cases)/total number of cases ] × 100%.
Toronto clinical scoring system（TCSS） | Baseline, 3 weeks, 6 weeks, 10 weeks
  The scale is an assessment of foot sensation and has a total score of 19, divided into three sections: symptom score of 6, reflex score of 8 and sensory score of 5. Symptom score: 0 = absent, 1 = present; reflex score: 0 = normal, 1 = diminished, 2 = absent; sensory score: 0 = normal, 1 = abnormal.
TCM syndromes efficacy score scale | Baseline, 3 weeks, 6 weeks, 10 weeks
  TCM syndromes efficacy score is 42, ranging from 0 (least severe) to 42 (most severe).
Regional temperatures of sole of the foot | Baseline, 6 weeks
  Before and after treatment, the temperature of the sole of the foot will be measured using an infrared thermal imager
Regional temperatures of instep | Baseline, 6 weeks
  Before and after treatment, the temperature of the instep will be measured using an infrared thermal imager
Regional temperatures of palm | Baseline, 6 weeks
  Before and after treatment, the regional temperature of the palm will be measured using an infrared thermal imager.
Regional temperatures of back of the hand | Baseline, 6 weeks
  Before and after treatment, the regional temperature of the back of the hand will be measured using an infrared thermal imager.
Patient Global Impression of Change(PGIC) | Baseline, 3 weeks, 6 weeks, 10 weeks
  PGIC is scored on a 7-point scale, with higher scores representing poorer efficacy. a score of 1 indicates that the subject perceives a great improvement in efficacy, 4 is no change before and after acupuncture treatment, and 7 is much worse after treatment.
Glycated haemoglobin (HbA1c） | Baseline, 6 weeks
Fasting blood glucose (FPG) | Baseline, 3 weeks, 6 weeks, 10 weeks
2-hour postprandial blood glucose (2hPG) | Baseline, 3 weeks, 6 weeks, 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D,M.D, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Li Y, Teng D, Shi X, Qin G, Qin Y, Quan H, Shi B, Sun H, Ba J, Chen B, Du J, He L, Lai X, Li Y, Chi H, Liao E, Liu C, Liu L, Tang X, Tong N, Wang G, Zhang JA, Wang Y, Xue Y, Yan L, Yang J, Yang L, Yao Y, Ye Z, Zhang Q, Zhang L, Zhu J, Zhu M, Ning G, Mu Y, Zhao J, Teng W, Shan Z. Prevalence of diabetes recorded in mainland China using 2018 diagnostic criteria from the American Diabetes Association: national cross sectional study. BMJ. 2020 Apr 28;369:m997. doi: 10.1136/bmj.m997. PMID 32345662
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Iqbal Z, Azmi S, Yadav R, Ferdousi M, Kumar M, Cuthbertson DJ, Lim J, Malik RA, Alam U. Diabetic Peripheral Neuropathy: Epidemiology, Diagnosis, and Pharmacotherapy. Clin Ther. 2018 Jun;40(6):828-849. doi: 10.1016/j.clinthera.2018.04.001. Epub 2018 Apr 30. PMID 29709457
- [Background] Zhang R, Lao L, Ren K, Berman BM. Mechanisms of acupuncture-electroacupuncture on persistent pain. Anesthesiology. 2014 Feb;120(2):482-503. doi: 10.1097/ALN.0000000000000101. PMID 24322588
- [Background] Dimitrova A, Murchison C, Oken B. Acupuncture for the Treatment of Peripheral Neuropathy: A Systematic Review and Meta-Analysis. J Altern Complement Med. 2017 Mar;23(3):164-179. doi: 10.1089/acm.2016.0155. Epub 2017 Jan 23. PMID 28112552
- [Background] Yu B, Li M, Huang H, Ma S, Huang K, Zhong Z, Yu S, Zhang L. Acupuncture treatment of diabetic peripheral neuropathy: An overview of systematic reviews. J Clin Pharm Ther. 2021 Jun;46(3):585-598. doi: 10.1111/jcpt.13351. Epub 2021 Jan 28. PMID 33511675
- [Background] He XF, Wei JJ, Shou SY, Fang JQ, Jiang YL. Effects of electroacupuncture at 2 and 100 Hz on rat type 2 diabetic neuropathic pain and hyperalgesia-related protein expression in the dorsal root ganglion. J Zhejiang Univ Sci B. 2017 Mar.;18(3):239-248. doi: 10.1631/jzus.B1600247. PMID 28271659
- [Derived] Luo N, Zeng YC, Fu BT, Low JW, Fang JQ. Investigating the Effectiveness of Electroacupuncture for Diabetic Peripheral Neuropathy and Exploring the Feasibility of Infrared Thermography as an Efficacy Assessment Tool: Study Protocol for a Randomized Controlled Trial. J Pain Res. 2024 Aug 23;17:2727-2739. doi: 10.2147/JPR.S472648. eCollection 2024. PMID 39193463